CLINICAL TRIAL: NCT01441076
Title: A Pilot Study of Anakinra in Behcet's Disease (BD)
Brief Title: Anakinra for Behcet s Disease
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 110241; 11-AR-0241 (Other: National Institute of Health)
Record Dates: First submitted 2011-09-24; First posted 2011-09-27 (Estimated); Results first posted 2017-05-12 (Actual); Last update posted 2017-05-12 (Actual); Status verified 2017-04

CONDITIONS: Autoimmune Connective Tissue Disorder; Immune System Diseases
Keywords: Behcet's Disease; Aphthous Ulcer; Uveitis; IL-1; Autoinflammation; BD
MeSH Terms: conditions — Immune System Diseases; Behcet Syndrome; Stomatitis, Aphthous; Uveitis | interventions — Interleukin 1 Receptor Antagonist Protein

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Anakinra (Experimental): Treatment with Anakinra 100mg subcutaneous daily with option to escalate dose up to 300mg subcutaneous daily
  Interventions: Drug: Anakinra

INTERVENTIONS:
Drug: Anakinra — Anakinra/Kineret[registered] is a recombinant, non-glycosylated form of the human interleukin-1 receptor antagonist (IL-1Ra)

SUMMARY:
Background:

- Behcet's disease (BD) is an autoimmune disease where the immune system attacks the body. People with BD may develop oral or genital ulcers, skin problems, and eye disease. Most drugs used to treat BD suppress the immune system, but they are not always helpful and may have side effects. A new drug, anakinra, may be able to treat BD with fewer side effects. Because it has not been studied in people with BD, anakinra is considered an experimental treatment.

Objectives:

- To test whether anakinra can be a safe and effective treatment for Behcet s disease.

Eligibility:

- People who have Behcet's disease with ongoing oral or genital ulcers for at least one month, or three or more flares of eye disease in the past 6 months.

Design:

* Participants will be screened with a physical exam and medical history. They will also have blood and urine tests. They will be divided into two groups: those with oral or genital ulcers and those with eye disease.
* All participants will keep a diary of symptoms for a month before starting the study drug.
* Participants with oral or genital ulcers will receive daily injections of anakinra for 3 to 6 months. Treatment will be monitored with frequent blood draws and daily diaries. Those who improve but do not have a full response to the drug may receive a higher dose. Those who improve after 6 months may have an extra 6 months on either anakinra or placebo to study the differences in response.
* Participants with eye disease will receive anakinra for up to 12 months. Treatment will be monitored with frequent blood draws, daily diaries, and regular eye exams.
* All participants will have a final study visit 1 month after stopping the study drug.

DETAILED DESCRIPTION:
Autoinflammatory diseases are illnesses characterized by episodes of inflammation that, unlike autoimmune disorders, lack the production of high titer autoantibodies or antigen-specific T cells. There is growing genetic and clinical evidence that Interleukin-1 (IL-1) plays a pathogenic role in several of these diseases. This exploratory study aims to examine the utility of anakinra in the treatment of adult subjects with Behcet s Disease (BD), a disease which shows similarities to the known anakinra-responsive autoinflammatory disorders, familial cold autoinflammatory syndrome (FCAS) and Muckle-Wells Syndrome (MWS). Anakinra is a recombinant form of the human interleukin-1 receptor antagonist that has been studied in rheumatoid arthritis (RA) and the autoinflammatory disorders. It has a half life of 4 to 6 hours with a FDA approved recommended dose of 100 mg/day subcutaneously for the treatment of rheumatoid arthritis.

This pilot study is designed to address: 1) the utility of anakinra in the treatment of BD; 2) the effect of anakinra on laboratory biomarkers in BD; and 3) an exploratory assessment of the safety of anakinra in individuals with Behcet's Disease.

Subjects with oral or genital ulcers will receive anakinra for three to six months. If five of the initial seven patients have a positive response, up to 20 patients with oral or genital ulcers will then be randomized to withdrawal or continuation of drug for six months once placebo is available. Patients with eye disease will be treated with anakinra for a total of twelve months without randomization to withdrawal. Clinical and biochemical correlates of inflammation will be measured at appropriate intervals to assess response and to further understand disease mechanisms.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Male or female subjects with BD associated inflammatory disease greater than or equal 18 years of age
  2. Participation in NIH study #03-AR-0173 ( Studies of the Natural History, Pathogenesis, and Outcome of Autoinflammatory Diseases )
  3. Diagnosis of Behcet s disease as determined by the International Study Group Criteria [17] or by complete Japanese Criteria [18].
  4. Active mucocutaneous disease as defined by at least one oral or genital ulcer within the past month.
  5. Stable dose of steroids, NSAIDs, DMARDs, or colchicine for four weeks prior to enrollment visit.
  6. For patients with ocular disease, no active intermediate or posterior disease at enrolment but history of an ocular flare (greater than or equal to 3 in the last 6 months) in the presence of any systemic anti-inflammatory therapy such as prednisone, azathioprine, Mycophenolate, methotrexate, cyclosporine, a tumor necrosis factor (TNF) inhibitor, or a combination of these medications. Patients must have developed active disease in the presence of at treatment with at least one of the following medications for at least six months: azathioprine, cyclosporine, or a TNF inhibitor.
  7. Females of childbearing potential (young women who have had at least one menstrual period regardless of age) must have a negative urine pregnancy test at screening and a negative serum pregnancy test at baseline prior to performance of any radiologic procedure or administration of study medication. Female patients will be screened for pregnancy at all NIH visits.
  8. Women of childbearing age and men able to father a child, who are sexually active, who agree to use a form of effective birth control, including abstinence.
  9. Either (1) a negative PPD test using 5 T.U. intradermal testing per Center for Disease Control and Prevention guidelines and no evidence of active tuberculosis (TB) on chest X-ray at the time of enrollment or (2) a positive PPD with no evidence of active TB by history or on chest X-ray at the time of enrollment and either past or present treatment with adequate therapy for at least one month prior to first dose of study medication. Full prophylaxis regimens will be completed. Subjects who have been Bacillus Calmette-Guerin (BCG)-vaccinated will also be skin-tested.
  10. Able to understand, and complete study-related questionnaires.
  11. Able and willing to give informed consent and abide with the study procedures.

EXCLUSION CRITERIA:

1. Treatment with a live virus vaccine during 3 months prior to baseline visit. No live vaccines will be allowed throughout the course of this study.
2. Patients with ocular disease who received local treatments other than eye drops (i.e. periocular or intraocular steroids, implants or other anti-inflammatory agents within 4 weeks prior to enrolment)
3. Current treatment with TNF inhibitors or discontinuation of TNF inhibitors within 8 weeks.
4. Presence of active infections or a history of pulmonary TB infection. Patients with a history of exposure to TB (positive PPD) who have not been treated with a TB prophylaxis regimen for at least one month.
5. Chest x-ray read by a radiologist with pleural scarring and/or calcified granuloma consistent with prior TB.
6. Positive test for or prior history of HIV, Hepatitis B or C.
7. History or concomitant diagnosis of congestive heart failure.
8. History of malignancy. Subjects deemed cured of superficial malignancies such as cutaneous basal or squamous cell carcinomas, or in situ cervical cancer may be enrolled.
9. Known hypersensitivity to Chinese Hamster Ovary (CHO) cell derived biologicals or any components of anakinra.
10. Presence of any additional rheumatic disease or significant systemic disease. For example, major chronic infectious/ inflammatory/ immunologic disease (such as inflammatory bowel disease, psoriatic arthritis, spondyloarthropathy, systemic lupus erythematosus in addition to autoinflammatory disease).
11. Presence of any of the following laboratory abnormalities at enrollment visit: creatinine > 1.5 times the upper limit of normal , white blood cell < 3.6 times10(9)/mm(3); platelet count < 75,000 mm(3); alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 2.0 times the upper limit of normal
12. Lactating females or pregnant females.
13. Subjects with asthma not adequately controlled on current inhaled therapy for at least four weeks.
14. Enrollment in any other investigational treatment study or use of an investigational agent, or has not yet completed at least 4 weeks or 5 half-lives, whichever is longer, since ending another investigational device or drug trial.
15. Subjects for whom there is concern about compliance with the protocol procedures.
16. Presence of other severe acute or chronic medical or psychiatric condition, or significant laboratory abnormality requiring further investigation that may cause undue risk for the subject s safety, inhibit protocol participation, or interfere with interpretation of study results, and in the judgment of the investigator would make the subject inappropriate for entry into this study.
17. Treatment within the past 12 months with canakinumab
18. Active neurologic disease which would require cyclophosphamide treatment. Active neurologic disease is defined as either new evidence of parenchymal (meningoencephalitis) or non-parenchymal (vascular complications including thrombosis) disease.
19. Subjects who experience an end organ flare after discontinuation of a TNF inhibitor as part of this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2011-09; Primary Completion 2014-10 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter C Grayson, M.D., Principal Investigator — National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aksentijevich I, Putnam CD, Remmers EF, Mueller JL, Le J, Kolodner RD, Moak Z, Chuang M, Austin F, Goldbach-Mansky R, Hoffman HM, Kastner DL. The clinical continuum of cryopyrinopathies: novel CIAS1 mutations in North American patients and a new cryopyrin model. Arthritis Rheum. 2007 Apr;56(4):1273-1285. doi: 10.1002/art.22491. PMID 17393462
- [Background] Aksentijevich I, Nowak M, Mallah M, Chae JJ, Watford WT, Hofmann SR, Stein L, Russo R, Goldsmith D, Dent P, Rosenberg HF, Austin F, Remmers EF, Balow JE Jr, Rosenzweig S, Komarow H, Shoham NG, Wood G, Jones J, Mangra N, Carrero H, Adams BS, Moore TL, Schikler K, Hoffman H, Lovell DJ, Lipnick R, Barron K, O'Shea JJ, Kastner DL, Goldbach-Mansky R. De novo CIAS1 mutations, cytokine activation, and evidence for genetic heterogeneity in patients with neonatal-onset multisystem inflammatory disease (NOMID): a new member of the expanding family of pyrin-associated autoinflammatory diseases. Arthritis Rheum. 2002 Dec;46(12):3340-8. doi: 10.1002/art.10688. PMID 12483741
- [Background] Feldmann J, Prieur AM, Quartier P, Berquin P, Certain S, Cortis E, Teillac-Hamel D, Fischer A, de Saint Basile G. Chronic infantile neurological cutaneous and articular syndrome is caused by mutations in CIAS1, a gene highly expressed in polymorphonuclear cells and chondrocytes. Am J Hum Genet. 2002 Jul;71(1):198-203. doi: 10.1086/341357. Epub 2002 May 24. PMID 12032915
- [Derived] Grayson PC, Yazici Y, Merideth M, Sen HN, Davis M, Novakovich E, Joyal E, Goldbach-Mansky R, Sibley CH. Treatment of mucocutaneous manifestations in Behcet's disease with anakinra: a pilot open-label study. Arthritis Res Ther. 2017 Mar 24;19(1):69. doi: 10.1186/s13075-017-1222-3. PMID 28335798

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Anakinra
Started | 6
Completed | 4
Not Completed | 2

BASELINE CHARACTERISTICS:
Arm/Group | Anakinra
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  LTE18 | 0
  BTWN | 6
  GTE65 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic | 0
  Not Hispanic or Latino | 6
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Hawaiian | 0
  Black | 1
  White | 4
  More than one race | 1
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Clinical Remission From Months 3-6
Description: Clinical remission was defined as no oral or vaginal ulcers on physical examination for 2 consecutive monthly visits from months 3-6.
Time Frame: Monthly study visits from months 3-6 during the trial
Population: Analysis included all subjects who enrolled in the trial, including those who terminated the study prior to month 6 due to perceived lack of efficacy of study drug.
Measure: Number; unit: Participants
Arm/Group | Anakinra
Number analyzed (Participants) | 6
Participants | 2

2. Secondary Outcome: Behcet's Disease Related Quality of Life (BDRQOL) Assessment Score
Description: The BDRQOL is a standardized assessment form in Behcet's disease composed of 30 items (answered true or not true) and each item is scored 0 or 1 (scoring range from 0 to 30). A total lower score indicates a better quality of life and a total higher score indicates a worse quality of life.
Time Frame: Month 6 study visit
Population: as for outcome 1
Measure: Median (Full Range); unit: Units on a scale
Arm/Group | Anakinra
Number analyzed (Participants) | 6
Units on a scale | 9.5 [0 to 22]

3. Secondary Outcome: Behcet's Syndrome Activity Scale (BSAS) Score
Description: The BSAS is a standardized assessment form in Behcet's disease. The BSAS score comprises 10 items. The total score possible is between 0-100. A total lower score indicates a less syndrome activity and a higher total score indicates more syndrome activity.
Time Frame: Month 6 study visit
Population: as for outcome 1
Measure: Median (Full Range); unit: Units on a scale
Arm/Group | Anakinra
Number analyzed (Participants) | 6
Units on a scale | 21.3 [0 to 44]

4. Secondary Outcome: Behcets Disease Current Activity Form (BDCAF) Score
Description: The BDCAF is a standardized assessment form in Behcet's disease to measure patient activity. Scoring is based on the history of new clinical features present over the preceding 4 weeks prior to assessment. The range of score is 0 - 12. A total lower score indicates less disease activity and a higher total score indicates more disease activity.
Time Frame: Month 6 study visit
Population: as for outcome 1
Measure: Median (Full Range); unit: Units on a scale
Arm/Group | Anakinra
Number analyzed (Participants) | 6
Units on a scale | 5 [4 to 6]

5. Secondary Outcome: Number of Genital Ulcers by Physician Evaluation
Description: Number of genital ulcers noted by physician evaluation
Time Frame: Month 6 study visit
Population: as for outcome 1
Measure: Median (Full Range); unit: genital ulcers in participants
Arm/Group | Anakinra
Number analyzed (Participants) | 6
genital ulcers in participants | 0 [0 to 0]

6. Secondary Outcome: Number of Oral Ulcers by Physician Evaluation
Description: Number of oral ulcers noted by physician evaluation
Time Frame: Month 6 study visit
Population: as for outcome 1
Measure: Median (Full Range); unit: oral ulcers in participants
Arm/Group | Anakinra
Number analyzed (Participants) | 6
oral ulcers in participants | 0.5 [0 to 2]

7. Secondary Outcome: Patient Global Score
Description: Global visual analogue scale taken by patients with a range of score of 0-100. Lower scores indicate least symptoms and higher scores indicate worst symptoms faced by the patient.
Time Frame: Month 6 study visit
Population: as for outcome 1
Measure: Median (Full Range); unit: Units on a scale
Arm/Group | Anakinra
Number analyzed (Participants) | 6
Units on a scale | 51.5 [3 to 91]

8. Secondary Outcome: Physician Global Score
Description: Global visual analogue scale administered by physicians with a range of score of 0-100. Lower scores indicate least symptoms and higher scores indicate worst symptoms faced by the patient.
Time Frame: Month 6 study visit
Population: as for outcome 1
Measure: Median (Full Range); unit: Units on a scale
Arm/Group | Anakinra
Number analyzed (Participants) | 6
Units on a scale | 8.5 [7 to 24]

9. Secondary Outcome: Behcet's Disease Related Quality of Life (BDRQOL) Assessment Score
Description: as for outcome 2
Time Frame: Baseline
Population: as for outcome 1
Measure: Median (Full Range); unit: Units on a scale
Arm/Group | Anakinra
Number analyzed (Participants) | 6
Units on a scale | 16 [10 to 24]

10. Secondary Outcome: Behcet's Syndrome Activity Scale (BSAS) Score
Description: as for outcome 3
Time Frame: Baseline
Population: as for outcome 1
Measure: Median (Full Range); unit: Units on a scale
Arm/Group | Anakinra
Number analyzed (Participants) | 6
Units on a scale | 46 [22 to 80.5]

11. Secondary Outcome: Behcets Disease Current Activity Form (BDCAF) Score
Description: as for outcome 4
Time Frame: Baseline
Population: as for outcome 1
Measure: Median (Full Range); unit: Units on a scale
Arm/Group | Anakinra
Number analyzed (Participants) | 6
Units on a scale | 6 [5 to 11]

12. Secondary Outcome: Number of Genital Ulcers by Physician Evaluation
Description: Number of genital ulcers noted by physician evaluation
Time Frame: Baseline
Population: as for outcome 1
Measure: Median (Full Range); unit: genital ulcers in participants
Arm/Group | Anakinra
Number analyzed (Participants) | 6
genital ulcers in participants | 0 [0 to 3]

13. Secondary Outcome: Number of Oral Ulcers by Physician Evaluation
Description: Number of oral ulcers noted by physician evaluation
Time Frame: Baseline
Population: as for outcome 1
Measure: Median (Full Range); unit: oral ulcers in participants
Arm/Group | Anakinra
Number analyzed (Participants) | 6
oral ulcers in participants | 3.5 [2 to 5]

14. Secondary Outcome: Patient Global Score
Description: as for outcome 7
Time Frame: Baseline
Population: as for outcome 1
Measure: Median (Full Range); unit: Units on a scale
Arm/Group | Anakinra
Number analyzed (Participants) | 6
Units on a scale | 73.5 [9 to 90]

15. Secondary Outcome: Physician Global Score
Description: as for outcome 8
Time Frame: Baseline
Population: as for outcome 1
Measure: Median (Full Range); unit: Units on a scale
Arm/Group | Anakinra
Number analyzed (Participants) | 6
Units on a scale | 16.5 [12 to 79]

ADVERSE EVENTS:
Groups:
- Anakinra: Treatment with Anakinra 100mg subcutaneous daily
Arm/Group | Anakinra
Serious Adverse Events (participants affected / at risk) | 1/6
Other Adverse Events (participants affected / at risk) | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Anakinra (N=6)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1
Presyncope (Nervous system disorders) | 1
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1
Thromboembolic event (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Anakinra (N=6)
Anemia (Blood and lymphatic system disorders) | 1
Blurred vision (Eye disorders) | 1
Eye disorders - Other, specify (Eye disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 2
Edema limbs (General disorders) | 2
Fatigue (General disorders) | 1
Allergic reaction (Immune system disorders) | 4
Bronchial Infection (Infections and infestations) | 1
Infections and infestations - Other, specify (Infections and infestations) | 1
Pharyngitis (Infections and infestations) | 1
Rhinitis infective (Infections and infestations) | 2
Upper respiratory infection (Infections and infestations) | 2
Vaginal infection (Infections and infestations) | 1
Vulval infection (Infections and infestations) | 1
Hypoglycemia (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Dizziness (Nervous system disorders) | 1
Mania (Psychiatric disorders) | 1
Urinary Frequency (Renal and urinary disorders) | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 2
Phlebitis (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No